CLINICAL TRIAL: NCT01265420
Title: The Efficacy and Safety of Xiaflex Injections for the Treatment of Thumb Cords in Dupuytren's Contractures
Brief Title: Efficacy and Safety of Xiaflex Injection for Treatment of Dupuytren's Contracture of the Thumb
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana Hand to Shoulder Center (Other)
Responsible Party: Principal Investigator, F. Thomas D. Kaplan, MD, MD, Indiana Hand to Shoulder Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHtSC-Thumb 101
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Dupuytren's Contracture
Keywords: Dupuytren; Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injectable clostridial collagenase (Experimental): Patients with thumb 1st web contracture secondary to Dupuytren's disease will be treated with 0.58mg of collagenase
  Interventions: Biological: Injectable clostridial collagenase

INTERVENTIONS:
Biological: Injectable clostridial collagenase — Injection of 0.58mg clostridial collagenase into Dupuytren's cord, up to three injections
  Other Names: Xiaflex

SUMMARY:
This study will evaluate the efficacy and safety of clostridial collagenase injections for treatment of Dupuytren's contracture of the thumb and first web space. The investigators hypothesis is that clostridial collagenase will have safety not significantly different to that demonstrated in Phase III clinical trials, and will be effective in significantly reducing the degree of thumb contracture.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (> 18 years) of either gender with an MP and/or IP joint contracture and a palpable cord of > 20 degrees of the thumb
* First web space contracture with a palpable cord due to Dupuytren's contracture

Exclusion Criteria:

* Prior surgical, percutaneous needle aponeurotomy or Xiaflex treatment for Dupuytren's contracture of the same thumb.
* Any subject using anti-coagulant therapy other than low dose aspirin (up to 150mg/day).
* Any subject in the opinion of the MD investigators with chronic, severe or terminal medical illness which would make them unsuitable for study participation.
* Any subject with known allergy to Xiaflex (Clostridial collagenase).
* Pregnant or nursing female
* Any subject who cannot conform to the study visit schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hand to Shoulder Center, Indianaplis, Indiana, United States

REFERENCES:
- [Background] Hurst LC, Badalamente MA, Hentz VR, Hotchkiss RN, Kaplan FT, Meals RA, Smith TM, Rodzvilla J; CORD I Study Group. Injectable collagenase clostridium histolyticum for Dupuytren's contracture. N Engl J Med. 2009 Sep 3;361(10):968-79. doi: 10.1056/NEJMoa0810866. PMID 19726771

RESULTS

PARTICIPANT FLOW:
Groups:
- Injectable Clostridial Collagenase: Patients were treated with 0.58 mg clostridial collagenase into palpable cord in 1st webspace
Period: Overall Study
Arm/Group | Injectable Clostridial Collagenase
Started | 7
Completed | 6 (One patient was seen at Day 10 but did not return for Day 30 evaluation)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Injectable Clostridial Collagenase
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 62 [55 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number Patients Obtaining Clinical Improvement (>50% Reduction in Contracture)
Time Frame: 30 days after last injection
Measure: Number; unit: participants
Arm/Group | Injectable Clostridial Collagenase
Number analyzed (Participants) | 6
participants
  >50% reduction in contracture | 5
  <50% reduction in contracture | 1

ADVERSE EVENTS:
Time Frame: Day 1 after injection to Day 30
Arm/Group | Injectable Clostridial Collagenase
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Injectable Clostridial Collagenase (N=7)
Ecchymosis (Skin and subcutaneous tissue disorders) | 7
Edema (Skin and subcutaneous tissue disorders) | 7
Pruritis (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
nausea (Gastrointestinal disorders) | 1
Skin Tear (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
1 patient was seen at Day 10, but not at day 30. At Day 10, patient met the primary endpoint

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No